CLINICAL TRIAL: NCT00072085
Title: Immunization Of Patients With Metastatic Melanoma Using A Recombinant GP100 Protein (184V) And A Class I Restricted Peptide From The GP100 Antigen
Brief Title: Immunization With gp100 Protein Vaccine in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000335441; NCI-03-C-0299; NCI-6210; NCT00069043 (obsolete NCT alias)
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2005-05

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; incomplete Freund's adjuvant

INTERVENTIONS:
Biological: aldesleukin
Biological: gp100 antigen
Biological: incomplete Freund's adjuvant

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells.

PURPOSE: This randomized phase II trial is studying immunization using two different gp100 protein vaccines to compare how well they work in treating patients with metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the clinical response in patients with metastatic melanoma immunized with recombinant gp100 protein (184V) emulsified in Montanide ISA-51 with or without gp100:209-217 (210M) peptide.

Secondary

* Compare the toxicity profile of these immunizations in these patients.

OUTLINE: This is a randomized study. Patients are assigned to 1 of 2 cohorts according to HLA-A2*0201 status. Patients assigned to cohort 1 are then randomized to 1 of 2 treatment arms.

* Cohort 1 (HLA-A2*0201-positive patients): Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive immunization comprising recombinant gp100 protein (184V) emulsified in Montanide ISA-51 subcutaneously (SC) on days 1, 22, 43, and 64 (1 course).
  * Arm II: Patients receive immunization comprising recombinant gp100 protein (184V) and gp100:209-217 (210M) peptide emulsified in Montanide ISA-51 SC on days 1, 22, 43, and 64 (1 course).
* Cohort 2 (HLA-A2*0201-negative patients): Patients receive immunization as in cohort 1, arm I.

In both cohorts, treatment continues in the absence of rapid disease progression or unacceptable toxicity.

In both cohorts, patients are evaluated 3-4 weeks after the fourth immunization. Patients achieving stable disease or a partial response receive retreatment according to their assigned cohort. Patients with progressive disease who are eligible for interleukin-2 (IL-2) receive retreatment according to their assigned cohort AND high-dose IL-2 IV over 15 minutes 3 times daily on days 2-5, 23-26, 44-47, and 65-68 (1 course). Patients receive up to 3 retreatment courses. Patients achieving a complete response (CR) receive 1 retreatment course beyond CR. Patients with progressive disease who are ineligible for IL-2 administration are removed from the study.

PROJECTED ACCRUAL: A total of 45-75 patients (30-50 for cohort 1 [15-25 per treatment arm] and 15-25 for cohort 2) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of metastatic melanoma
* Measurable disease
* Progressive disease during or after prior standard treatment with or without interleukin-2

PATIENT CHARACTERISTICS:

Age

* 16 and over

Performance status

* ECOG 0-2

Life expectancy

* More than 6 months

Hematopoietic

* WBC at least 3,000/mm^3
* Platelet count at least 90,000/mm^3
* Lymphocyte count greater than 500/mm^3

Hepatic

* Bilirubin no greater than 2.0 mg/dL (less than 3.0 mg/dL for patients with Gilbert's syndrome)
* ALT and AST less than 3 times normal
* Hepatitis B surface antigen negative

Renal

* Creatinine no greater than 2.0 mg/dL

Cardiovascular

* No symptomatic cardiac disease

Immunologic

* No active systemic infection
* No autoimmune disease
* No known immunodeficiency disease
* No known hypersensitivity to study agents
* No form of primary or secondary immunodeficiency
* No opportunistic infection
* HIV negative

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* No prior gp100 peptide vaccine

Chemotherapy

* More than 6 weeks since prior nitrosoureas

Endocrine therapy

* No concurrent systemic steroid therapy

Radiotherapy

* Not specified

Surgery

* Prior recent (within the past 3 weeks) minor surgical procedures allowed

Other

* Recovered from prior therapy (toxicity no greater than grade 1)
* More than 3 weeks since prior systemic anticancer therapy
* No other concurrent systemic anticancer therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-09; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Principal Investigator — NCI - Surgery Branch
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland